CLINICAL TRIAL: NCT00261053
Title: A Phase II Exploratory, Open-label Study of the Safety and Efficacy of Recombinant Human C1 Inhibitor for the Treatment of Acute Attacks in Patients With Hereditary Angioedema
Brief Title: Recombinant Human C1 Inhibitor for the Treatment of Acute Attacks in Patients With Hereditary Angioedema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharming Technologies B.V. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1 1202-01
Record Dates: First submitted 2005-12-01; First posted 2005-12-02 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Genetic Disorders
MeSH Terms: conditions — Genetic Diseases, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Open-label i.v. administration of 100 U/kg rhC1INH
  Interventions: Drug: i.v. recombinant human C1 inhibitor

INTERVENTIONS:
Drug: i.v. recombinant human C1 inhibitor

SUMMARY:
The purpose of this single-center study is to explore the efficacy, safety, tolerability and pharmacokinetics/pharmacodynamics of recombinant human C1 inhibitor in the treatment of acute attacks in patients with hereditary angioedema.

ELIGIBILITY:
Main inclusion Criteria:

* Clinical and laboratory diagnosis of HAE
* Plasma level of functional C1INH of less than 50% of normal
* Severe attack of abdominal, facial-oro-pharyngeal, genito-urinary and/or peripheral HAE.

Main exclusion Criteria:

* Acquired angioedema
* Pregnancy or breastfeeding
* Participation in another clinical study within prior 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2003-06; Primary Completion 2005-09 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Primary outcomes: Relief of angioedema symptoms

SECONDARY OUTCOMES:
Secondary outcomes: Safety and tolerability; pharmacokinetics/pharmacodynamics

CONTACTS AND LOCATIONS:
Overall Officials: Jan Nuijens, MD, PhD, Study Chair — Pharming Technologies B.V.
Locations (1):
- For information contact Sonja Visscher, Leiden, Netherlands